CLINICAL TRIAL: NCT02895958
Title: Open Label Study of the Safety and Efficacy of FDC Zepatier (Elbasvir+Grazoprevir +/- Ribavirin)Administered in a Community Based Setting to HCV Infected G1/4 Treatment naïve Patients on Stable Opiate Substitution Therapy With Cirrhotic and Non-cirrhotic Liver Disease
Brief Title: The Dublin Zepatier Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient study participants enrolled
Sponsor: Mater Misericordiae University Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Jack Lambert, Infectious Diseases Consultant, Mater Misericordiae University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEP-HEPC-001
Record Dates: First submitted 2016-08-30; First posted 2016-09-12 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of Zepatier (Other)
  Interventions: Drug: Zepatier

INTERVENTIONS:
Drug: Zepatier — Zepatier (elbasvir and grazoprevir +/- Ribavirin) will be administered in a community setting to HCV infected G1/4 treatment naïve patients on stable opiate substitution therapy with Cirrhotic and Non-cirrhotic liver disease

SUMMARY:
Evaluation of Zepatier in a community-based setting among cirrhotic and non-cirrhotic patients on stable opiate substitution therapy.

DETAILED DESCRIPTION:
Hard-to-reach groups such as those attending addiction and homeless services are particularly at risk for HCV-associated liver disease progression as they do not engage in treatment, have poor attendance records for appointments, and are at risk of progression to cirrhosis without evaluation and detection. These patients are therefore "silently" progressing in the community and may be close to decompensation. Once a patient goes over that critical stage from compensated to decompensated cirrhosis, the cost to the patient in terms of their health, and the cost to the state in terms of the management of cirrhosis related complications are great.

As part of this investigator-led community-based treatment protocol we aim to demonstrate the utility of an integrated community-based care partnership between primary and secondary care to best evaluate and treat such hard to reach populations.

We aim to actively find fibrosis levels of HCV related liver disease using the FibroScan diagnostic tool, and support patients to be treated for their HCV with the newly available DAAs and be cured of their HCV infection and disease through:

1. Active case finding by travelling to the services used by 'at risk' groups as opposed to giving appointments to the patient to attend hospital.
2. Locating HCV patients (with positive RNA or HCV antigen) that are 'lost to follow up'.
3. Staging and risk-stratifying HCV patients locally to support access to therapy.
4. Educating HCV patients around new assessment tools and treatments.
5. Setting up and supporting the initiation of treatment in the community e.g. daily dispensing of medication/treatment with methadone.
6. Providing on-going harm reduction advice on preventing reinfection.
7. Work in partnership with Methadone prescribing GP practices and Drug Treatment Centres from the North and South Dublin catchment area

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject must be HCV treatment naive. Subject is willing and able to understand and provide written informed consent prior to participation in this study.
3. Documented chronic HCV infection (RNA positive), HCV RNA levels > 10x4 IU/ml.
4. Documented HCV genotype 1 and 4.
5. Documented HIV and HBV uninfected (HIV Ab negative, HBsAg negative)
6. A female is eligible to enter and participate in the study if she is of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
   * Child-bearing potential, has a negative pregnancy test (serum β-HCG) at screen and agrees to an acceptable barrier and/or hormonal method of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the approved product label and the instructions of a physician): Sterilization (female subject or male partner of female subject). Male and female subjects must agree to 7 months post-treatment contraception if taking ribavirin and one month post- treatment contraception for Zepatier only.
7. Stable attender in the site of enrolment (receiving OST at least 3 months before enrolment and were at least 80 % adherent to OST appointments)
8. Venous access available for blood monitoring.
9. Fibroscan done as per HSE Hepatitis C Advisory Group guidelines.
10. Safety bloods done prior to study including a HGB > 9.5g/dL, platelets > 75,000, AST < 10x ULN, albumin levels > 30g/L.

Exclusion Criteria:

1. 1. Child Pugh B or C (see Appendix 10.1 for Child-Pugh Classification)
2. HCV non-G1/G4
3. History of decompensated liver disease
4. Laboratory exclusions include platelet count <75,000, albumin <30gm/L, Alanine aminotransferase (ALT) >10 times the upper limit of normal (ULN).
5. Subject is enrolled in one or more investigational drug protocols, which may impact on assessment of HCV treatment with Zepatier (+/-ribavirin).
6. Subject is, in the opinion of the investigator, unable to complete the study dosing period and protocol evaluations and assessments.
7. Patients with alcohol and drug use problems that in the view of investigator will compromise adherence to compliance with the study will be excluded.
8. Subject is either pregnant or breastfeeding.
9. Subject suffers from any serious medical condition (such as pancreatitis, diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction), which in the opinion of the Investigator, would compromise the safety of the subject.
10. Subject has a pre-existing mental, physical, or substance abuse disorder that, in the opinion of the Investigator, may interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments.
11. Subject has a history of inflammatory bowel disease or intestinal malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction, which, in the opinion of the Investigator, may interfere with drug absorption or render the subject unable to take oral medication.
12. Subject has any acute laboratory abnormality at screening, which, in the opinion of the Investigator, would preclude the subject's participation in the study of an investigational compound. If subjects are found to have an acute Grade 4 laboratory abnormality at screening, this test may be repeated once within the 45-day screening window. Any verified Grade 4 laboratory abnormality would exclude a subject from study participation.
13. Subject has received treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to Screening, or has an anticipated need for these agents within the study period.
14. Subjects who require treatment with any contraindicated medications (as outlined in the SPC) within 14 days of commencement of investigational product, or an anticipated need during the study.
15. Subject has a history of allergy to any of the treatment products or any excipients therein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Sustained viral response (SVR) against HCV at 12 weeks after treatment | 12 weeks post-treatment

SECONDARY OUTCOMES:
Sustained viral response (SVR) against HCV at 24 weeks after completion of study treatment | 24 weeks post-treatment
Incidence of adverse events during course of treatment | Weeks 0-16 of treatment
Characteristics of adverse events | Week -8 pre-treatment to Week 24 post treatment
Incidence of treatment discontinuation over course of treatment | Weeks 0-16 of treatment
Rates of premature discontinuation of drug for clinical or laboratory reasons | Weeks 0-16 of treatment
Evaluation of percentage relapse at 12 and 24 weeks post treatment | weeks 12 and 24 post treatment
Percentage of re-infection as evaluated by repeat HCV RNA positivity at weeks 12 and 24 post-treatment | Weeks 12 and 24 post-treatment
Safety and feasibility of model of community based integrated care with community dispensation and supervision of DAA therapy to treat 'hard to reach' HCV infected patients | End of study
Change of quality of life assessment questionnaire score (EQ-5D-5L) administered at baseline, 12 weeks, and 24 weeks post-treatment | End of study

CONTACTS AND LOCATIONS:
Locations (1):
- Thompson Centre, Dublin, Ireland